CLINICAL TRIAL: NCT05041543
Title: A Randomized, Double-blinded, Placebo-controlled, Dose Escalation, Phase 1 Clinical Trial to Evaluate the Safety and Tolerability of NTX-101 in Healthy Volunteers
Brief Title: Safety and Tolerability of NTX-101 in Korean Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pinotbio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTX-101-P1
Record Dates: First submitted 2021-08-24; First posted 2021-09-13 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers
Keywords: Ophthalmic Solutions; Eye Drops; Eye Diseases; Ischemic Optic Neuropathy; Glaucoma
MeSH Terms: conditions — Eye Diseases; Optic Neuropathy, Ischemic; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- NTX-101 Group A (Experimental): Day 1: One time administration, single drop. 4 subjects randomized 3:1 to NTX-101 or placebo.
  Interventions: Drug: NTX-101; Drug: Placebo
- NTX-101 Group B (Experimental): Day 1: One time administration, single drop. Day 3-7: Two time administration, one drop each time (12 hours apart). Total 9 times administration. 8 subjects randomized 6:2 to NTX-101 or placebo.
  Interventions: Drug: NTX-101; Drug: Placebo
- NTX-101 Group C (Experimental): Day 1: One time administration, single drop. Day 3-7: Two time administration, one drop each time (12 hours apart). Total 9 times administration. 8 subjects randomized 6:2 to NTX-101 or placebo.
  Interventions: Drug: NTX-101; Drug: Placebo
- NTX-101 Group D (Experimental): Day 1: One time administration, two drops. Day 3-7: Two time administration, two drops each time (12 hours apart). Total 9 times administration. 8 subjects randomized 6:2 to NTX-101 or placebo.
  Interventions: Drug: NTX-101; Drug: Placebo
- NTX-101 Group E (Experimental): Day 1: One time administration, four drops. Day 3-7: Two time administration, four drop each time (12 hours apart). Total 9 times administration. 8 subjects randomized 6:2 to NTX-101 or placebo.
  Interventions: Drug: NTX-101; Drug: Placebo

INTERVENTIONS:
Drug: NTX-101 — Eye drops, topical administration
Drug: Placebo — Placebo as eye drops

SUMMARY:
A double-blinded, placebo controlled, multiple dose, randomized, single site, phase 1 clinical trial to evaluate safety, tolerability, and pharmacokinetics of NTX-101 topical eye drop in Korean healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects who have voluntarily agreed to the participation of this study upon sufficient explanation of the purpose, procedure, and the characteristics of the experimental drug of the trial prior to participation
2. Subjects of ages between 19 and 45 years inclusive and with Body Mass Index (BMI) between 18.0 and 27.0

Exclusion Criteria:

1. Clinical History

   * Subjects with a clinically significant history of the gastrointestinal, hepatic, cardiovascular, pulmonary, endocrine, renal, urological, immunologic, musculoskeletal, neurological, psychiatric, hematological, ocular, otolaryngologic disorder not deemed acceptable by the PI
   * Subjects with a clinically significant history of disorder that can affect the experimental drug's absorption, distribution, metabolism, and excretion (e.g. Crohn's disease, peptic ulcer, surgery to stomach and intestine (excluding appendectomy and herniorrhaphy)) not deemed acceptable by the PI
2. Ocular History

   * Subjects with a suspected history or symptoms of visual organ disorder, including keratitis, uveitis, retinitis, dry eye syndrome, and strabismus.
   * Subjects with corrected visual acuity of below 20/40 (0.5 in Han Chun Suk chart)
   * Subjects with history of ocular surgery, excluding those who received laser eye surgery 6 months prior to screening
   * Subjects who have experienced complications from wearing contact lens, used contact lens in the past month, or cannot adhere to the prohibition of using contact lens during the study
   * Subjects with other anomalies discovered at the ocular examination upon screening
3. Clinical Examination

   * Subjects with a resting blood pressure of >140 mmHg or <90 mmHg diastolic, >90 mmHg or <60 mmHg systolic, or heartrate exceeding 100 per minute
   * Subjects with inadequate levels of the following criteria upon repeated examination

     1. AST or ALT >1.25 x upper limit of normal level
     2. Total bilirubin >1.5 x upper limit of normal
     3. eGFR level from CKD-EPI equation < 90 mL/min/1.73m²
     4. Positive blood serum result (HBsAg, HCV Ab, HIV Ab, Syphilis reagin test)
   * Subjects who show anomalies or have the following results repeatedly in the electrocardiogram (including, but not limited to, major arrhythmia, multifocal PVC, 2° A-V block anomaly, etc.)

     1. PR interval ≥ 210msec
     2. QRS complex ≥ 120msec
     3. QTcF interval ≥ 450msec
4. Allergy, Hypersensitivity, or Substance Abuse

   * Subjects with hypersensitivity to the components or additives of the experimental drug
   * Subjects with clinically significant allergy (excluding mild allergic rhinitis that does not require medication) or prior history of hypersensitivity to other drugs (aspirin, antibiotics, etc.)
   * Subject with history of substance abuse (especially drugs that act on Central Nervous System, such as sedatives, Central Nervous System depressants, opioids, or psychotropic drugs, etc.) or positive result from screening test (methamphetamine, marijuana, opium, cocaine, amphetamine, ecstasy)
5. Prohibited drug/food

   * Subjects who have taken drug metabolism stimulator or suppressor within 1 month of the first experimental drug administration
   * Subjects who have received vaccination within 8 weeks prior to the first experimental drug administration or is expecting to receive before the end of study
   * Subjects who have taken prescribed medicine (including prescribed herbal medicine) 14 days prior or over-the-counter drugs (including vitamin supplements) 10 days prior to the administration of the experimental drugs that may affect the study determined by the PI
   * Subjects who have taken within 7 days prior to the first administration of the experimental drug or cannot stop taking food that may affect the drug's absorption, distribution, metabolism, and excretion (e.g. grapefruit juice, garlic extract, broccoli, kale, etc.)
   * Subjects who have participated in other pharmacokinetic or other clinical studies and have taken experimental drugs 6 months prior to this study
6. Blood Donation and Transfusion

   * Subjects who have donated whole blood within 2 months prior to the first administration of the experimental drug or have donated blood components within 1 month prior to the administration of the experimental drug
   * Subjects who have received blood transfusion within 1 month prior to the administration of the experimental drug
7. Contraceptives

   * Subjects who use inadequate contraceptives during the study that have not been clinically accepted

     1. Use of intrauterine device that have been proved to prevent pregnancy
     2. Use of condoms (male or female) with spermicide
     3. Vasectomy
     4. Tubal ligation or hysterectomy
     5. Sperm donation during the study period
8. Others

   * Subjects who refuses to stop taking xanthine-containing food from 3 days prior to the first administration of the experimental drug until the end of study (e.g. coffee, green tea, black tea, cola, cocoa, chocolate, energy drinks, etc.)
   * Subjects who refuses to stop drinking excessive alcohol (>30 g/day) from 3 days prior to the first administration of the experimental drug until the end of study
   * Subjects who refuses to stop smoking during the hospitalization period
   * Subjects deemed unfit for this study by the Principal Investigator

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation: Incidence, type, and severity of Adverse Events (AE) | 7 Days

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum plasma concentration (Cmax) | Pre-dose, 15, 30, 45 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours after first and last administration
Pharmacokinetics (PK): Area under the curve (AUC) | Pre-dose, 15, 30, 45 minutes, 1, 2, 3, 4, 6, 8, 12, 24 hours after first and last administration

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea